CLINICAL TRIAL: NCT06402370
Title: Amyloid PET in Patients With Mild Cognitive Impairment and Early Dementia
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0444
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: MCI
MeSH Terms: interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET scan — [18F]Vizamyl

SUMMARY:
The National Institute on Aging together with the Alzheimer's Association (NIA-AA) recently proposed the ATN classification which is based upon the pathological processes present in Alzheimer's disease (amyloid, tau and neurodegeneration). The amyloid and tau status can be defined using cerebrospinal fluid analysis but also non-invasively using an amyloid or tau PET scan. The N status can be defined using an [18F]-FDG PET scan which is in Belgium part of standard of care. Recently, it has been demonstrated, using different amyloid PET tracers, that early-frame amyloid scans can be a surrogate for [18F]-FDG PET scan.

DETAILED DESCRIPTION:
With the general aging of the population, neurodegenerative diseases such as Alzheimer have an increasing prevalence. Recently, anti-β-amyloid-antibodies such as aducanumab and donanemab are under development. These treatments urge for techniques allowing early diagnosis and treatment monitoring during disease. [18F]FDG PET allows the visualization of metabolic disturbances and aid in the early diagnosis of Alzheimer, Amyloid PET is able to detect the amyloid plaques which can be present years before symptom onset. A recent meta-analysis demonstrated that amyloid PET has a high sensitivity (0.91) and specificity (0.81) in the differential diagnosis between Alzheimer and controls, however very poor specificity (0.41) was observed when differentiating between Alzheimer and patients with mild cognitive impairment.

The National Institute on Aging together with the Alzheimer's Association (NIA-AA) recently proposed the ATN classification which is based upon the pathological processes present in Alzheimer's disease (amyloid, tau and neurodegeneration). The amyloid and tau status can be obtained using cerebrospinal fluid analysis but also non-invasively using an amyloid or tau PET scan. The N status can be obtained using an [18F]FDG PET scan which is in Belgium part of standard of care. Both the [18F]FDG PET scan and the amyloid scans using [18F]Vizamyl are also proposed in the diagnostic algorithm for early and differential diagnoses of dementia .

Perfusion scans using [15O]H2O have shown a good correlation with [18F]FDG PET, illustrating the potential of perfusion as a proxy for neuronal dysfunction. Previously, it has been demonstrated that early amyloid scans represent perfusion and can therefore be used as a proxy for neuronal activity.

Next generation PET/CT scanners, such as the Omni Legend have a very high sensitivity which may enable ultra-short PET scans, which is important is this vulnerable patient group, or dynamic scans with a high effective time resolution due to the possibility to acquire short time frames with reasonable noise characteristics. Moreover, the ultrashort scan may limit the movement artefacts frequently encountered in this study population.

The investigators hypothesize that a one minute scan 5 minutes postinjection is sufficient to determine the N-status of a patients and that a one minute scan 90-110 minutes postinjection can determine the A-status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild cognitive impairment or early stage dementia who have a MRI and [18F]FDG PET/CT scan as part of routine clinical work-up

Exclusion Criteria:

* Patient is not able to understand the study Patient is not able to lie still in the scanner for at least 30 minutes Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with early Alzheimer and mild cognitive impairment
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
N-status | 2 years
  N-status can be determined using ultrashort early frame amyloid scans of 1 minute
A-status | 2 years
  A-status can be determined with a one minute scan 60-90 minutes after injection

CONTACTS AND LOCATIONS:
Overall Officials: Donatienne Van Weehaeghe, MD PhD, Principal Investigator — UZ Gent
Locations (1):
- Van Weehaeghe D, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No